CLINICAL TRIAL: NCT03569384
Title: Feasibility & Effect of a Tele-rehabilitation Program for Chronic Obstructive Pulmonary Disease vs. Standard Rehabilitation
Acronym: TELEKOL-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Eurostars (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-TELE KOL 1
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: The study is a prospective randomized controlled trial comparing the effects of tele-rehabilitation and conventional rehabilitation in patients with COPD.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group "tele-rehabilitation" (Experimental): Video Consultation (VC) Sessions: Each patient will have the opportunity to have minimum one VC per week the first month, one VC each second week the second month one VC a month Retraining breath: Patients will also be instructed to use different techniques to breath during the video consultations with the physiotherapist. Chat Sessions: Each patient has the opportunity to chat with the physiotherapist any time via the chat module of the system. Workout Sessions with a Virtual Physiotherapist Agent (VPA):
  The patient will train according to what is decided by the physiotherapist and the patient in the VC or chat meetings. Normally, the patients will train 10-20 minutes daily at home with its individual and tailored VPA. Patients' security: In order to minimize the risks of possible accidents while performing the exercises, the patient will answer questions before and after each exercise performance that the physiotherapist can follow in real time.
  Interventions: Combination Product: Tele Rehab
- Control (Active Comparator): COPD patients in the control group will undergo the conventional standardized rehabilitation program as implemented at the Department of Respiratory Medicine and Allergy, Aarhus University Hospital. The program is an 8 weeks program consisting of 2 weekly group training sessions at the hospital with instruction by a physiotherapists and 6 hours of education about COPD and its treatment.
  Interventions: Combination Product: Tele Rehab

INTERVENTIONS:
Combination Product: Tele Rehab — The intervention group will obtain telerehabilitation

SUMMARY:
Introduction In order to guarantee chronic patients and elderly a high quality service from health care organizations in the coming decades, new technologies have been implemented to treat patients from a distance. There is still a need for more studies on the efficacy and cost-effectiveness of tele-rehabilitation (TR) and its long-term effects needs also to be determined. To guarantee individuals with chronic obstructive pulmonary diseases (COPD) a high quality service from health care organizations in the coming decades and economically save the national health systems for an expensive bill for the treatment of COPD, new actions plans has to be taken into use. Hereby, more patients can be treated with less human resources while still sustaining or even improving today's services. The importance of such welfare action plans has to maintain a high quality of service that individuals with COPD are willing to accept. Here, TR seems to be a good welfare action plans. Despite proof of improved cost-effectiveness, no studies support the benefits of TR in COPD patient with respect to adherence, security, treatment efficacy and improved quality of life.

Aim To assess and compare the feasibility and effect of a tele-rehabilitation program with a new and innovative TR platform (NITRP) compared to standard treatment with respect to exercise capacity, quality of life and activities of daily living in patients with COPD.

Method and material The study is a prospective randomized controlled trial comparing the effects of tele-rehabilitation and conventional rehabilitation in patients with severe COPD. 54 patients fulfilling the inclusion criteria will be randomized in two groups to either a 8 week tele-rehabilitation program or a conventional COPD rehabilitation program at the hospital. Participants will be tested at baseline, 8 weeks, 3 and 6 months after cessation of the training programs. In the intervention group, a real- and a virtual physiotherapist agent will facilitate the rehabilitation.

Ethical considerations This study will not pose any risk to the patient as compared to current practice. Participation is voluntary and the patient may at any time withdraw from the study without consequences for future care or treatment. The questionnaires and the test methods used are clinically recognized instruments. Signed informed consent will be obtained from the all participants after verbal and written information and before the study starts. The study will not be initiated before approval from the Ethics Committee and the Data Protection Agency has been obtained. The study will follow the general research ethical rules as expressed in the Helsinki Declaration II.

DETAILED DESCRIPTION:
Introduction

To guarantee chronic patients and elderly a high quality service from health care organizations in the coming decades, new technologies has been implemented to treat patients from a distance. This document reflects the latest research studies based on tele-rehabilitation (TR), its application in chronic lung diseases and the topics that still needs to be investigated.

Tele-rehabilitation Studies of TR in patients with lymphedema (Galiano-Castillo et al., 2014) or COPD (Paneroni et al., 2014)(Tousignant et al., 2012)(Dinesen, Seeman, and Gustafsson, 2011)(Dinesen, Huniche, and Toft, 2013) or in the orthopedic areas as, lower back (Palacín-Marín, Esteban-Moreno, Olea, Herrera-Viedma, & Arroyo-Morales, 2013), knee (Cabana et al., 2010) (Tousignant, Moffet, et al., 2011) (Tousignant, Boissy, et al., 2011) and shoulder (Eriksson, Lindström, Gard, & Lysholm, 2009)(Eriksson, Lindström, & Ekenberg, 2011) show that tele-technology has been developed to a level where it is possible to treat, test and follow-up patients from a distance. Patients who have not been offered such solutions face increased risks of hospital-acquired infections (Dancer, 2009) and longer travel and waiting time to get treated. The public sector expects higher expenditure due to treatment and transportation cost, specifically in chronic patients and the elderly whose numbers tends to increase according to demographics trend (Palacín-Marín et al., 2013)(Barros, Francisco, Zanchetta, & César, 2011)(Parker & Thorslund, 2007)(Yach, Hawkes, Gould, and Hofman, 2004). Such facts points to the need of creating and improving solutions that overcome such health care challenges.

TR seems to be a good approach to reach patients in low inhabited areas (Hill and Sppath, 2010), changing health care to self-care (Haarder, 2011), empowering patient's awareness of their disease and increasing the flexibility patients need to acquire to obtain healthier behaviors. Although the interest in TR research is high, there is still a need for more studies on the efficacy (Paneroni et al., 2014) and cost-effectiveness of TR (Paneroni et al., 2014) (Langberg, Lindahl, Kidholm, and Dinesen, 2014) just as the long-term effects of TR have to be determined (Langberg et al., 2014).

Chronic obstructive pulmonary disease (COPD) COPD is among the most resource costly diseases we face in our century (Kjøller, Juel, and Kamper-Jørgensen, 2007). In Denmark, approximately 430,000 people have COPD of which around 50,000 have severe COPD (Kirkegaard N, Brandt A, Timm H, 2013)(Mannino, Doherty, and Sonia Buist, 2006). Eriksen (Eriksen and Vestbo, 2010) states that up to 42.3% of patients with COPD discharged from hospitals are readmitted the following year, and 17% of patients treated in emergency departments require hospitalization. Danish pulmonary physicians concluded that COPD cost the Danish society three billion DKK in 2002 (Hos, 2007) where up to 20% of the most severe COPD patients consume over 70% of the total health expenditure (Jansson et al., 2002). Nowadays, some municipalities have already problems with offering rehabilitation services to all COPD patients in some areas in Denmark (Kjøller et al., 2007). Actions implementing TR for COPD patients have been started and research begins to show some improvements.

Pulmonary rehabilitation in COPD The objective of treatment for patients with COPD is to delay the progression of the disease, prevent acute exacerbations, improve quality of life, reduce symptoms and reduce mortality. Rehabilitation of COPD includes among others physical training and patient education (Sundhedsstyrelsen, 2007). There is a need for an improved prevention and treatment of exacerbations (Barnes, Calverley, Kaplan, & Rabe, 2013). Despite the poor evidence about determinants of physical activity and impact of treatment in COPD patients (Gimeno-Santos et al., 2014), a wide range of interventions are commonly used by physiotherapist to treat individuals with COPD (Kozu et al., 2011),(Kenn, Gloeckl, and Behr, 2013) (Garrod and Lasserson, 2007). Researchers have shown significant improvement in general condition (Lacasse, Guyatt, and Goldstein, 1997)(Ries, Kaplan, Limberg, and Prewitt, 1995)(Lacasse, Goldstein, Tj, and Martin, 2009)(Nava, 1998)(Simpson, Killian, McCartney, Stubbing, and Jones, 1992), quality of life (Wijkstra et al., 1995)(Bendstrup 1997), long-term survival (Godoy 2007), sputum clearance (Garrod 2007) (Oldenburg 1979); Health-related quality of life (Almagro 2013) (Blackstock 2013) (Jones, 2013)(Bendstrup et al. 1997), training of muscle strength and exercise tolerance (Ortega et al., 2002)(Bendstrup et al., 1997), walking distance (Ries et al. 2007) (Ringbaek 2008) (Wedzicha et al., 1998), exercise capacity, endurance (Lacasse et al., 1997) (Ries et al., 1995) (Lacasse et al., 2009) (Nava 1998) (Simpson et al., 1992); days of hospitalization (Ries et al., 2007) (Griffiths et al., 2000), tachypnea (Lacasse et al., 1997) (Ortega et al., 2002) and morbidity (Godoy, 2007). Although the advantages of PR are many, its implementation should be placed alongside the routine treatment options (Ozalevli 2010). It has been shown that the frequency of emergency department presentations and hospital admissions in COPD patients was significantly reduced after participation in early discharge care with ongoing follow-up support (Lawlor et al., 2009).

Tele-rehabilitation in COPD Tele-rehabilitation at home is feasible and well accepted by patients, although technology may be perceived as difficult (Paneroni et al., 2014)(Tousignant et al., 2012). It seems to improve walking capacity, dyspnea, quality of life and daily physical activity (Paneroni et al., 2014). The interaction between the COPD patients at home and the healthcare professionals at the clinic through TR has evolved as a dialogue channel forming the basis for mutual learning processes and new relationships (Dinesen 2011). Here, patients exhibit four types of attitudes about their tele-rehabilitation: indifference, learning as part of situations in everyday life, feeling of security and motivation for performing physical training (Dinesen et al., 2013). Preliminary evaluations from tele-rehabilitation initiatives in Scotland showed tele-rehabilitation to be more cost effective for patients living in remote areas compared to an out-reach- or centralized model (Hill 2010).

Conclusion There is still a need for more studies of the efficacy and cost-effectiveness of TR, just as also the long-term effects of TR have to be determined. To guarantee individuals with COPD a qualitative service from health care organizations in the coming decades and economically save the national health systems for an expensive bill to treating COPD, new actions plans has to be taken in mind in order to treat more patients with less human resources and still sustaining or improving today's services. The importance of such welfare action plans has to maintain a quality of service that individuals with COPD are willing to accept. Here, TR seems to be a good welfare action plans. Despite improved cost effectiveness, evidence supporting patient ´s adherence and security, treatment efficacy and improvements of quality of life with tele-rehabilitation in COPD is still warranted.

Aim To assess and compare the feasibility and effect of a tele-rehabilitation program with a new and innovative TR platform (NITRP) compared to standard COPD rehabilitation with respect to exercise capacity, quality of life and activities of daily living in patients with COPD.

The primary purpose of the study is to assess the effect of tele-rehabilitation with a NITRP compared to standard COPD rehabilitation on exercise capacity and quality of life in COPD patients based on the following hypotheses:

Activities of daily living, exercise capacity and health-related quality of life are equal or improved by tele-rehabilitation compared to conventional COPD rehabilitation.

The secondary purpose is to investigate the efficacy and cost effectiveness of tele-rehabilitation with a NITRP compared to standard COPD rehabilitation on "number of acute exacerbations and number of visits to the health care system in a period of time" and "rehabilitation- and transportation costs" in rehabilitation of COPD patients based on the following hypothesis:

The rehabilitation costs of tele-rehabilitation are lower or equal compared to conventional rehabilitation.

METHOD AND MATERIAL

Design:

The study is a prospective randomized controlled trial comparing the effects of tele-rehabilitation and conventional rehabilitation in patients with COPD.

Patients 54 adult patients with moderate to severe COPD referred for conventional COPD rehabilitation in the outpatient clinic at the Department of Respiratory Medicine and Allergy, Aarhus University Hospital

Inclusion criteria

In order to be eligible to participate in this study, the patient must meet all of the following criteria:

A diagnosis of COPD (FEV1/FVC < 70% in a stable phase of the disease) Age > 18 years Referred for conventional COPD rehabilitation Compliant patient willing to fulfill the study requirements Signed informed consent Oxygen therapy is not an obstacle for participation.

Exclusion criteria

A potential patient who meets any of the following criteria will be excluded from participation in this study if:

Musculoskeletal disorders limiting training Dizziness, significant sensory or motor disabilities, dementia or terminal malignant disease precluding training Severe comorbidities such as i.e. unstable heart disease, dysregulated diabetes, known malignant disease, any other illness making the patient inappropriate for participating in the study Non-compliant patient Severe vision or hearing impairment Non-Danish speaking Unwillingness or inability to follow the protocol COPD exacerbation in the preceding 6 weeks

Sample size calculation In this non-inferiority study of tele-rehabilitation vs. standard rehabilitation, we will use 6MWT as the primary outcome. Power calculations based on previous rehabilitation studies in COPD results I 54 patients that should participate in this study. The biggest allowed difference in 6MWT: +/- 35 m (Puhan et al 2008) to accept the H0: same mean difference, assuming equal group sizes, means that 18 patients is needed in each group. A drop-out rate less than or equal to 30% is expected (Sohanpal et al 2012). The maximum dropout rate in the present study is set to 40%. Thus, the final power calculations results in 54 patients, significance rate 0.05. Therefore, 27 patients will enrolled in each group.

Recruitment All COPD patients referred for rehabilitation at the Department of Respiratory Medicine and Allergy, Aarhus University Hospital that might be eligible will be informed about the study by their respiratory physician or physiotherapist when evaluated after referral for rehabilitation. The patients will be asked if they are interested in participating in this study, and if so, they will receive verbal and written information. An enrolment letter will also be hung up at the outpatient clinic to inform potential participants about the project. An advertisement will be published in local newspapers, on AUH facebook and on www.forsoegsperson.dk (Appendix 4). In this information the study is explained in detail. Potential participants are entitled to at least one day consideration time before they decide whether to participate in the trial. They have the right to be accompanied by a family member, friend or acquaintance for the oral information they will receive previous to the enrolment. . The patients have to give their informed signed consent to the principal investigator or his designee before the patient can enter the trial. Clinical stability will be assessed by the physician. If patients are eligible they will be randomized to the intervention group or control group.

Treatment of subjects There will be no changes in the patients' regular treatment due to participation in the tele-rehabilitation study.

Investigational treatment The intervention is the use of a tele-rehabilitation program during 8 weeks. The patient's training time will be registered automatically. The control group will receive standard COPD rehabilitation.

Escape medication In case of a COPD exacerbation or any other medical incidence, the patient will be treated to the discretion of the clinician in charge and excluded from the study. However, the patients will be offered to be included again at the moment clinical stability is reached and the patient again fulfils inclusion criteria.

Randomisation, blinding & treatment allocation Randomisation will allocate patients to either the intervention or control group and will be performed electronically.

Study procedures The trial is registered in the public database of Clinical Trials.gov. After informed consent, the patients will be screened at baseline and physical examination, pulmonary function tests and 6MWT will be performed.

Information on comorbidities and smoking status will be registered. All patients will be asked to fill in the questionnaires on health-related quality of life, general-well-being and anxiety. Patients will be asked to wear a pedometer and record steps during 7 days and will be instructed not to change their daily routine while wearing this device. After returning back the pedometer, patients allocated to the intervention group will receive instructions about the tele-rehabilitation program while patients allocated to the control group will start the standard rehabilitation program.

In week 8, the intervention group will again receive a pedometer to register steps for 7 days during the intervention. 8 weeks after the end of the intervention program, pulmonary function tests, 6MWT and the questionnaires will be repeated. The same investigations and questionnaires are performed at follow-up after 3 and 6 months after the end of the rehabilitation program.

Patients allocated to the control group will follow the same procedure during the first 9 weeks, except not using tele-rehabilitation.

Control group COPD patients in the control group will undergo the conventional standardized rehabilitation program as implemented at the Department of Respiratory Medicine and Allergy, Aarhus University Hospital. The program is an 8 weeks program consisting of 2 weekly group training sessions at the hospital with instruction by a physiotherapists and 6 hours of education about COPD and its treatment.

Intervention group The intervention group will follow this procedure Video Consultation (VC) Sessions: Each patient will have the opportunity to have minimum one VC per week the first month, one VC each second week the second month one VC a month the rest of the trial. Here the physiotherapist, via history will extract the information needed to calibrate the daily tele rehabilitation program according to patient's physical status and needs.

Retraining breath: Patients will also be instructed to use different techniques to breath during the video consultations with the physiotherapist. The patient receives advice on how to the use breathing retraining techniques such as pursed lip breathing. Because COPD patients suffer from obstructed airways, the goal for them using PLB will be to increase their positive expiratory pressure.

Chat Sessions: Each patient has the opportunity to chat with the physiotherapist any time via the chat module of the system. The patient and physiotherapist will be reminded via mail, anytime someone is writing in the chat, allowing the users to interact when needed.

Workout Sessions with a Virtual Physiotherapist Agent (VPA): The patient will train according to what is decided by the physiotherapist and the patient in the VC or chat meetings. Normally, the patients will train 10-20 minutes daily at home with its individual and tailored VPA. Instead of ergometer bike training, the patient will receive some easy training tools such as elastics and weights that can be used in the different exercises showed by the VPA to reach the same intensity of work out. The VPA will then be animated to motivate and encourage the patient to exercises at home. A digital diary will automatically register the data obtained by the system on patient's performance.

Patients' security: In order to minimize the risks of possible accidents while performing the exercises, the patient will answer questions before and after each exercise performance that the physiotherapist can follow in real time via scales and use to calibrate the performance of the virtual physiotherapist. The patient has the opportunity to chat with the physiotherapist 24 hours per day any time if needed and for consultation reasons.

Study parameters/endpoints

Primary endpoint:

Change in the 6MWT measured at week 9.

Secondary endpoint:

Change in the 6MWT measured 3 and 6 months after cessation of the tele-rehabilitation program compared to baseline.

Change in total score in health-related quality of life measured by SGRQ at week 9, and 3 and 6 months after cessation of the tele-rehabilitation program compared to baseline.

Change in total score in health-related quality of life measured by GAD-7 at week 9, and 3 and 6 months after cessation of the tele-rehabilitation program compared to baseline.

Change in component scores (symptoms, activity & impact) in health-related quality of life measured by SGRQ at week 9, and 3 and 6 months after cessation of the tele-rehabilitation program compared to baseline.

Cost of the tele-rehabilitation program

End point measures

Pulmonary function tests (PFT):

PFT are done as part of the routine follow-up and performed to prove disease stability. The following pulmonary function indices will be registered:

Forced expiratory volume in 1 second (FEV1) Forced vital capacity (FVC)

6 minute walk test A 6 minute walk test will be performed at baseline, after 8 weeks, and after 3 and 6 months after cessation of the program to assess exercise performance. The purpose of this test is to see how far and fast the test person can walk during 6 minutes. This test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. During this test the patient will be asked to walk between two cones placed 30 meters apart. The patient is asked to go to the speed he thinks he can walk without stopping during 6 minutes. Oximetry, pulse and Borgs Dyspnea Score are tracked before, after 6, 7, and 8 minutes. Total distance is recorded after 6 minutes. The patient stops walking after 6 minutes but recovery is also recorded at 7 and 8 minutes.

Pedometer:

To assess the physical activity status of the patient, measurement of the number of steps walked is an indication of the magnitude of physical activity. In controlled laboratory settings, the Yamax Digi-walker SW-200 has consistently been shown to be among the most accurate. It's a small device worn on the belt or waist and responds to vertical accelerations of the hip during gait cycles.

Questionnaires:

At baseline, and after 8 weeks, 3 and 6 months, the patient will be asked to self-administer the following questionnaires on quality of life and general well-being:

IADL Instrumental Activity of Daily Living consists of seven questions related to shopping, housework, cooking, walks, money management, handling of medications and use of telephone. Both patients and their closest relatives (mostly spouses) should reply. For each of the seven questions, a score of zero indicates no need for help, one indicates some needs and two indicates inability to perform an activity without assistance. A total score is calculated on a scale from 0 to 14. Higher scores indicate greater dependence. The form has been translated into Danish (Appendix 1), SGRQ Sct. Georges Respiratory Questionnaire is a disease specific, self-administered questionnaire with 50 items comprising two domains with 3 components as symptoms, activity and impacts. Each is scored from 0-100, with higher scores corresponding to worse health related quality of life. SGRQ has been developed for COPD patients and found to be a valid measure of health related quality of life (Appendix 2).

GAD-7:

The General Anxiety Disorder Score measures the presence and severity of general anxiety disorder. It is a 7 self-rated items. Each item scores 0-3. The total score range is 0-21. Reliability and validity are excellent (Appendix 3).

COPD exacerbations The number of exacerbations and visits to the general practitioner, emergency room or hospital during rehabilitation and follow-up will be registered, first via a diary and corroborated then by short interviews performed during follow-up at 8 weeks and 3 and 6 months after cessation of training.

Cost The average cost of the hospital rehabilitation program and transportation per patients for an eight weeks standard and tele-rehabilitation program and transportation will be calculated.

Data Collection Information about patient demographics, lung function (spirometry with measurement of FEV1 and FVC), oxygen saturation, comorbidities, smoking habits, BMI, blood pressure, visits to the clinic, number of exacerbations, use of any public health care service and cost of it will be registered at each visit.

Data analysis There will be used Wilcoxon rank sum test for assessing, the primary endpoint comparing the performance of the physical functions tests between the intervention group and control group from base line to 8 weeks, 3 and 6 months after and for the test variables with correction for multiple comparisons. A p-value less than 0.05 will be considered statistically significant. All patients will be analyzed in the groups they originally were randomized from according to the intention-to-treat principles.

Differences in activities of daily living and health-related quality of life between the two groups from baseline to 8 weeks, 3 and 6 months after will be compared with Chi2 test or Fischer's exact test for categorical data. Continuous data will be compared with t -tests or Wilcoxon rank sum test depending on distribution. A p-value less than 0.05 will be considered statistically significant.

Copyrights, distribution and implications Authorship must meet the Vancouver rules, and everyone who has contributed under this framework will be named in the author list. The authors will try to publish the results of the study in international peer-reviewed journals and present them at relevant conferences. Moreover, the results will be published in other relevant media. All positive, negative and inconclusive results will be published

Ethical issues Since rehabilitation is a standard treatment offer, it is not expected that this study will result in any risk to patients. Participation is voluntary and the patient may, at any time, withdraw from the study without consequences for future care or treatment. Questionnaires and test methods used are clinically recognized instruments. An informed written consent will be obtained from the participants after verbal and written information. The Regional Research Ethics Committee will be applied in order to obtain their consent to carry out the study. The is approved by the Data Protection Agency for permission for data recording and storage of data. The data will be rendered anonymous through a code system and stored safely in accordance with applicable rules of the organizers. The study follows the general research ethics rules as expressed in the Helsinki Declaration II ("World Medical Association Declaration of Helsinki: Ethical Principles for Medical Research involving Human Subjects," 2000).

Passed on information from the patient journal system Patient data as mentioned below will be passed on from the electronic patient files to the project.

Gender, age, marital status, comorbidities and smoking status will be passed on at the beginning of the study to compare the data at the end of the trial.

Telephone number, address and or E-mail from participants in the focus group will be passed on with the goal to contact the participant in the case there is a break in the connection via the tele rehab devices or if we need to send a new updated devices.

Health status, number of exacerbations in the last period, days of hospitalization, number of visits to the hospital or number of visits from healthcare suppliers to participants at home will be used to calculate the health care expenditure for each participant.

Economy MD, Ph.D. Elisabeth Bendstrup, MD Anders Løkke, MD, ph.d. Ole Hilberg and physiotherapist José Cerdan has initiated this project and sought various foundations to execute this study.

Elisabeth Bendstrup, Anders Løkke and Ole Hilberg are the responsibles of the investigation for this study and have no financial ties to the donors.

The study is predominantly financed by EURO STARS Foundation (1,500,000 kr.) and Aarhus University (about 450,000 kr.).

Physio R & D, Laster Technologies, Cortrium and bookBeo are providing the the technology, network, hardware, software and support needed for free.

Aarhus University Hospital provides locations and resources as needed and pays for the costs of the control group training. Aarhus University Hospital is also responsible for the administration and disbursement of funding.

Enrolled participants do not receive honorees for participating in this study. Transport costs associated with the trial will be covered by Aarhus University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of COPD (FEV1/FVC < 70% in a stable phase of the disease)
* Age > 18 years
* Referred for conventional COPD rehabilitation
* Compliant patient willing to fulfill the study requirements
* Signed informed consent (Oxygen therapy is not an obstacle for participation).

Exclusion Criteria:

* Musculoskeletal disorders limiting training
* Dizziness, significant sensory or motor disabilities, dementia or terminal malignant disease precluding training
* Severe comorbidities such as i.e. unstable heart disease, dysregulated diabetes, known malignant disease, any other illness making the patient inappropriate for participating in the study
* Non-compliant patient
* Severe vision or hearing impairment
* Non-Danish speaking
* Unwillingness or inability to follow the protocol
* COPD exacerbation in the preceding 6 weeks

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-03-30 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
6 Minutes Walk Test | 9 weeks
  Change in the 6MWT measured at week 9

SECONDARY OUTCOMES:
6 Minutes Walk Test | 3 and 6 months after cessation of the tele-rehabilitation program
  Change in the 6MWT measured 3 and 6 months after cessation of the tele-rehabilitation program compared to baseline
Health-related quality of life SGRQ (in total score) | at week 9, and 3 and 6 months after cessation of the tele-rehabilitation program
  Change in total score in health-related quality of life measured by SGRQ at week 9, and 3 and 6 months after cessation of the tele-rehabilitation program compared to baseline.
Health-related quality of life GAD-7 | at week 9, and 3 and 6 months after cessation of the tele-rehabilitation program
  Change in total score in health-related quality of life measured by GAD-7 at week 9, and 3 and 6 months after cessation of the tele-rehabilitation program compared to baseline.
Health-related quality of life SGRQ (symptoms, activity & impact) | at week 9, and 3 and 6 months after cessation of the tele-rehabilitation program
  Change in component scores (symptoms, activity & impact) in health-related quality of life measured by SGRQ at week 9, and 3 and 6 months after cessation of the tele-rehabilitation program compared to baseline.
Cost of the tele-rehabilitation program | at week 9
  Cost of the tele-rehabilitation program

CONTACTS AND LOCATIONS:
Overall Officials: Jose Cerdan, PhD student, Principal Investigator — Aarhus University Hospital
Locations (1):
- Jose Cerdan, Århus C, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
The study is approved by the Data Protection Agency for permission for data recording and storage of data. The data will be rendered anonymous through a code system and stored safely in accordance with applicable rules of the organizers. The study follows the general research ethics rules as expressed in the Helsinki Declaration II ('World Medical Association Declaration of Helsinki: Ethical Principles for Medical Research involving Human Subjects', 2000).

REFERENCES:
- [Result] Tsai LL, McNamara RJ, Moddel C, Alison JA, McKenzie DK, McKeough ZJ. Home-based telerehabilitation via real-time videoconferencing improves endurance exercise capacity in patients with COPD: The randomized controlled TeleR Study. Respirology. 2017 May;22(4):699-707. doi: 10.1111/resp.12966. Epub 2016 Dec 19. PMID 27992099
- [Result] Zanaboni P, Dinesen B, Hjalmarsen A, Hoaas H, Holland AE, Oliveira CC, Wootton R. Long-term integrated telerehabilitation of COPD Patients: a multicentre randomised controlled trial (iTrain). BMC Pulm Med. 2016 Aug 22;16(1):126. doi: 10.1186/s12890-016-0288-z. PMID 27549782
- [Derived] Cross AJ, Thomas D, Liang J, Abramson MJ, George J, Zairina E. Educational interventions for health professionals managing chronic obstructive pulmonary disease in primary care. Cochrane Database Syst Rev. 2022 May 6;5(5):CD012652. doi: 10.1002/14651858.CD012652.pub2. PMID 35514131
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633
- See also: Telerehab platform we use — http://optimov.com